CLINICAL TRIAL: NCT03917381
Title: First-in-human, Open-label, Dose-escalation Trial With Expansion Cohorts to Evaluate Safety of GEN1046 in Subjects With Malignant Solid Tumors
Brief Title: GEN1046 Safety Trial in Patients With Malignant Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1046-01; 2018-003402-63 (EudraCT Number); MOH_2019-05-08_006011 (Registry Identifier: Clinical Research Site - mytrial); 2023-509059-15 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2019-04-11; First posted 2019-04-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Docetaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): Acasunlimab will be administered as monotherapy.
  Interventions: Biological: Acasunlimab
- Expansion (Experimental): Acasunlimab will be administered as monotherapy or in combination with either docetaxel, pembrolizumab, or pembrolizumab + standard chemotherapy in separate expansion cohorts.
  Interventions: Biological: Acasunlimab; Biological: Acasunlimab in combination with docetaxel (in a single expansion cohort); Biological: Acasunlimab in combination with pembrolizumab (in a separate expansion cohort); Biological: Acasunlimab in combination with pembrolizumab and standard chemotherapy (in separate expansion cohorts)

INTERVENTIONS:
Biological: Acasunlimab — Acasunlimab will be administered intravenously once every 21 days (in selected expansion cohorts acasunlimab will be administered intravenously once every 21 days for the first 2 cycles, and every 42 days in subsequent cycles).
  Other Names: GEN1046; DuoBody®-PD-L1x4-1BB
Biological: Acasunlimab in combination with docetaxel (in a single expansion cohort) — Acasunlimab and docetaxel will be administered intravenously once every 21 days.
  Other Names: GEN1046; DuoBody®-PD-L1x4-1BB
  Arms: Expansion
Biological: Acasunlimab in combination with pembrolizumab (in a separate expansion cohort) — Acasunlimab and pembrolizumab will be administered intravenously once every 21 days or every 42 days, respectively.
  Other Names: GEN1046; DuoBody®-PD-L1x4-1BB
  Arms: Expansion
Biological: Acasunlimab in combination with pembrolizumab and standard chemotherapy (in separate expansion cohorts) — Acasunlimab and pembrolizumab and standard chemotherapy will be administered intravenously once every 21 days for 4 cycles, followed by treatment with acasunlimab and pembrolizumab once every 21 days.
  Other Names: GEN1046; DuoBody®-PD-L1x4-1BB
  Arms: Expansion

SUMMARY:
The goal of this trial is to learn about the antibody acasunlimab (an antibody also known as GEN1046) when it is used alone and when it is used together with standard of care treatment (docetaxel) or another antibody cancer drug, pembrolizumab (with or without chemotherapy), for treatment of patients with certain types of cancer. All subjects will receive active drug; no one will receive placebo.

This trial has 2 parts. The purpose of the first part is to find out if acasunlimab at various doses is safe and to find out the best doses of acasunlimab to use. The purpose of the second part is to give acasunlimab to more subjects to see how well the doses of acasunlimab selected in the first part work against cancer when given alone and how well they work when given with pembrolizumab with or without chemotherapy.

Trial details include:

* The average trial duration for an individual subject will be about 74 weeks.
* The average treatment duration for an individual subject will be about 21 weeks.
* The visit frequency will be weekly at first and lessening over time until visits are only once every 3 weeks.

DETAILED DESCRIPTION:
The trial is an open-label, multi-center safety trial of acasunlimab (GEN1046). The trial consists of 2 consecutive parts: a first-in-human (FIH) dose escalation (phase 1) and an expansion (phase 2a). The expansion part of the trial will be initiated once the Recommended Phase 2 Dose (RP2D) has been determined.

ELIGIBILITY:
Key Inclusion Criteria:

For Dose Escalation:

• Have a histologically or cytologically confirmed non-CNS solid tumor that is metastatic or unresectable and for whom there is no available standard therapy

For Expansion:

• Have histologically or cytological confirmed diagnosis of relapsed or refractory, advanced and/or metastatic NSCLC, EC, UC, TNBC, SCCHN, or cervical cancer who are not anymore candidates for standard therapy For separate expansion cohorts: metastatic NSCLC without prior systemic treatment regimens for metastatic disease.

For Both Dose Escalation and Expansion

* Have measurable disease according to RECIST 1.1
* Have Eastern Cooperative Oncology Group (ECOG) 0-1
* Have an acceptable hematological status
* Have acceptable liver function
* Have an acceptable coagulation status
* Have acceptable renal function

Key Exclusion Criteria:

* Have uncontrolled intercurrent illness, including but not limited to:

  * Ongoing or active infection requiring intravenous treatment with anti-infective therapy, or any ongoing systemic inflammatory condition requiring further diagnostic work-up or management during screening.
  * Symptomatic congestive heart failure (Grade III or IV as classified by the New York Heart Association), unstable angina pectoris or cardiac arrhythmia
  * Uncontrolled hypertension defined as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg, despite optimal medical management
  * Ongoing or recent evidence of autoimmune disease
  * History of irAEs that led to prior checkpoint treatment discontinuation
  * Prior history of myositis, Guillain-Barré syndrome, or myasthenia gravis of any grade
  * History of chronic liver disease or evidence of hepatic cirrhosis
  * History of non-infectious pneumonitis that has required steroids or currently has pneumonitis
  * History of organ allograft (except for corneal transplant) or autologous or allogeneic bone marrow transplant, or stem cell rescue within 3 months prior to the first dose of acasunlimab
  * Serious, non-healing wound, skin ulcer (of any grade), or bone fracture
* Any history of intracerebral arteriovenous malformation, cerebral aneurysm, new (younger than 6 months) or progressive brain metastases or stroke
* Prior therapy:

  * Radiotherapy within 14 days prior to first dose of acasunlimab. Note: palliative radiotherapy will be allowed.
  * Treatment with an anti-cancer agent (within 28 days or after at least 5 half-lives of the drug, whichever is shorter), prior to acasunlimab administration. Accepted exceptions are bisphosphonates (e.g., pamidronate, zoledronic acid, etc.) and denosumab
* Toxicities from previous anti-cancer therapies that have not adequately resolved

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Number of Participants With Dose Limiting Toxicity (DLT) | During first cycle (21 days) for each cohort
  Toxicities will be graded for severity according to Common Terminology Criteria for Adverse Events (CTCAE) criteria version 5.0.
Dose Escalation and Monotherapy Expansion Cohorts: Number of Participants With Adverse Events (AEs) | From first dose until the end of the study (up to 60 days after the last dose)
Expansion Cohort 1: Objective Response Rate (ORR) | Up to 3 years
  ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) based on response evaluation criteria in solid tumours (RECIST).

SECONDARY OUTCOMES:
Expansion Cohort 1: Number of Participants With AEs | From first dose until the end of the study (up to 60 days after the last dose)
Combination Therapy Expansion Cohorts: Number of Participants With AEs | From first dose until the end of the study (up to 60 days after the last dose)
All Parts: Area Under the Concentration-Time Curve from Time Zero to Last Quantifiable Concentration (AUClast) of GEN1046 | Predose and postdose at multiple timepoints up to end of safety follow up (up to 60 days after last dose)
All Parts: Maximum Observed Plasma Concentration (Cmax) of GEN1046 | Predose and postdose at multiple timepoints up to end of safety follow up (up to 60 days after last dose)
All Parts: Number of Participants with Anti-drug Antibodies (ADAs) | Up to 3 years
  Venous blood samples will be collected for measurement of serum concentrations of ADAs.
Dose Escalation and Expansion Cohorts 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13: ORR | Up to 3 years
  ORR is defined as the percentage of participants with BOR of CR or PR based on RECIST v1.1.
Dose Escalation and Expansion Cohorts 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13: Disease Control Rate (DCR) | Up to 3 years
  The DCR is defined as the percentage of participants with confirmed BOR of CR, PR, or Stable Disease (SD) according to RECIST v1.1.
All Parts: Duration of Response (DoR) | Up to 3 years
  DOR is defined as the time from first documentation of response (CR or PR) to the date of the first documented progression or death whichever occurs earlier based on RECIST v1.1.
Expansion Cohort 1: Progression Free Survival (PFS) | Up to 3 years
  PFS is defined as the number of days from Day 1 in Cycle 1 to the first documented progression or death due to any cause, whichever occurs first based on RECIST version 1.1.
Expansion Cohort 1: Overall survival (OS) | Up to 3 years
  OS is defined as the number of days from Day 1 in Cycle 1 to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (57):
- United States (14):
  - Mayo Clinic, Phoenix, Arizona
  - Yale University Cancer Center, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - University of Iowa Hospitals, Iowa City, Iowa
  - Norton Healthcare Inc, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone, New York, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Levine Cancer Institute, Atrium Health, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - University Hospital Brno, Brno
  - Nemocnice AGEL Ostrava-Vítkovice a.s., Nový Jičín
  - Fakultni nemocnice Olomouc, Olomouc
- Georgia (4):
  - High Technology Hospital Medcenter, Batumi
  - LLC "TIM - Tbilisi Institute of Medicine", Tbilisi
  - LTD Consilium Medulla, Tbilisi
  - Tbilisi State Medical University and Ingorovka High Medical Technology University Clinic Ltd, Tbilisi
- Hungary (3):
  - Onkologiai Klinika, Debrecen
  - BKMK Hospital, Kecskemét
  - Pulmonology Hospital Törökbálinti, Törökbálint
- Israel (4):
  - Rambam Health Care Campus RHCC - Rambam Medical Center, Haifa
  - Hadassah Medical Organization HMO - Sharett Institute of Oncology, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Ramat Gan, Tel Litwinsky
- Italy (8):
  - Policlinico San'Orsola, Bologna
  - IRCCS - Istituto Europeo di Oncologia IEO, Milan
  - Istituto Nazionale Tumori - Fondazione Pascale Italy, Napoli
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - AUSL Romagno-Ravenna, Ravenna
  - Policlinico Uni. Campus Bio-Medico, Roma
  - Regina Elena National Cancer Institute, Rome
  - ASST Sette Laghi "Ospedale di Circolo e Fondazione Macchi ", Varese
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Medpolonia Sp. z o.o., Poznan
  - Specialist Hospital in Prabuty, Prabuty
  - Dom Lekarski SA, Szczecin
  - Maria Sklodowska Curie National Research Instutute of Oncology, Warsaw
- Spain (11):
  - Hospital Universitario Vall dHebron, Barcelona
  - IOB-Hospital Quironsalud Barcelona, Barcelona
  - START Madrid-FJD, Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - START Madrid-CIOCC, Madrid
  - NEXT Oncology Madrid, Madrid
  - Hospital Universitario La Princesa, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Clinico De Valencia, Valencia
- Turkey (Türkiye) (3):
  - Gulhane Training and Research Hospital, Ankara
  - Trakya University Hospital, Edirne
  - Medical Point Izmir Hospital, Karşıyaka
- ARENSIA Exploratory Medicine LLC, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muik A, Garralda E, Altintas I, Gieseke F, Geva R, Ben-Ami E, Maurice-Dror C, Calvo E, LoRusso PM, Alonso G, Rodriguez-Ruiz ME, Schoedel KB, Blum JM, Sanger B, Salcedo TW, Burm SM, Stanganello E, Verzijl D, Vascotto F, Sette A, Quinkhardt J, Plantinga TS, Toker A, van den Brink EN, Fereshteh M, Diken M, Satijn D, Kreiter S, Breij ECW, Bajaj G, Lagkadinou E, Sasser K, Tureci O, Forssmann U, Ahmadi T, Sahin U, Jure-Kunkel M, Melero I. Preclinical Characterization and Phase I Trial Results of a Bispecific Antibody Targeting PD-L1 and 4-1BB (GEN1046) in Patients with Advanced Refractory Solid Tumors. Cancer Discov. 2022 May 2;12(5):1248-1265. doi: 10.1158/2159-8290.CD-21-1345. PMID 35176764